CLINICAL TRIAL: NCT04516005
Title: Effect of Foot Reflexology on Blood Pressure and Pulse Rate: A Randomized Clinical Trial in Stage-2 Hypertensive Patients
Brief Title: Effect of Foot Reflexology on Blood Pressure and Pulse Rate: A Randomized Clinical Trial
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Khon Kaen University (Other)
Responsible Party: Principal Investigator, Praew Kotruchin, Assistant professor, Khon Kaen University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: HE611181
Record Dates: First submitted 2020-08-10; First posted 2020-08-17 (Actual); Last update posted 2020-08-17 (Actual); Status verified 2020-08

CONDITIONS: Reflexology, Hypertension, Acupressure, Traditional Medicine
Keywords: hypertension; reflexology; acupressure; traditional medicine
MeSH Terms: conditions — Hypertension

STUDY DESIGN:
Intervention Model Description: a single-center randomized clinical trial
Who Masked: Investigator
Masking Description: The statistical analysis investigator was blinded to the randomization group
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- foot reflexology (Experimental): Foot reflexology was performed in every participant in the foot reflexology group after resting for 5 minutes in a sitting position by the same researcher who was trained and certified by the Department of Thai Traditional and Alternative Medicine, Ministry of Health.
  Interventions: Procedure: foot reflexology
- control (No Intervention): The control group received conventional treatment including anti-HT medications according to the standard HT guideline's recommendations. In the end of the follow-up visit, every participants were informed to adhere to their medication and were encouraged to have healthy lifestyles including salt restriction, regular exercise, and consuming healthy diets.

INTERVENTIONS:
Procedure: foot reflexology — Acupressure was applied at the plantar side of the right foot at the first metatarsal bone, around 1-1.5 centimeters proximal to the first metatarsophalangeal joint. (Figure 2) Approximately 3-kilogram pressure was applied by using a knuckle of the right index finger (dorsal part of the proximal interphalangeal joint in flexing position) in a perpendicular manner and held for 15 seconds (sec) then released for 5 sec. This hold-release cycle was done 5 times over the course of 2 min. This method was recommended by the Department of Thai Traditional and Alternative Medicine in accordance with the Zone theory and the Meridian theory.
  Arms: foot reflexology

SUMMARY:
Hypertension (HT) has been known for its prominent risk of cardiovascular events. Although there are various pharmacological choices, many patients fail to adhere with them. Therefore, adjunctive non-pharmacological treatment is a promising approach. Foot Reflexology is one of a complementary therapies that has been proved for its ability to decrease blood pressure (BP), however, there is limited data in patients with stage-2 HT. We aimed to examine the effectiveness of foot reflexology as adjunctive therapy for BP lowering. This was a single-center randomized clinical trial. Hypertensive patients who were regularly followed up at the hypertension clinic were enrolled and randomized into the intervention group (n=47) and control group (n=47). Foot reflexology was performed in the intervention group during a clinical visit. Office BP and pulse rate (PR) were measured before and immediately at 15 minutes (min) and 30 min after the procedure in the intervention group and after resting in the control group.

DETAILED DESCRIPTION:
Background Hypertension (HT) has been known for its prominent risk of cardiovascular events. Although there are various pharmacological choices, many patients fail to adhere to them. Therefore, adjunctive non-pharmacological treatment is a promising approach. Foot Reflexology is one of the complementary therapies that has been proved for its ability to decrease blood pressure (BP), however, there is limited data in patients with stage-2 HT.

Objective To examine the effectiveness of foot reflexology as adjunctive therapy for BP lowering.

Methods This was a single-center randomized clinical trial. Hypertensive patients who were regularly followed up at the hypertension clinic were enrolled and randomized into the intervention group (n=47) and control group (n=47). Foot reflexology was performed in the intervention group during a clinical visit. Office BP and pulse rate (PR) were measured before and immediately at 15 minutes (min) and 30 min after the procedure in the intervention group and after resting in the control group.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosed stage-2 HT (defined by office SBP≥140 mmHg and/or DBP ≥90 mmHg at first hospital visit)
* On stable anti-HT drugs for at least 3 months before enrollment.

Exclusion Criteria:

* Pregnant women
* History of foot surgery or bone fracture
* Skin disease of the foot
* Diabetes neuropathy

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 94 (Actual)
Dates: Start 2015-11-01 (Actual); Primary Completion 2016-05-31 (Actual); Study Completion 2016-10-31 (Actual)

PRIMARY OUTCOMES:
Change of blood pressure level | Change from Baseline Systolic Blood Pressure at 15 minutes
  The office blood pressures (BP) were measured by a nurse at baseline and at 15 and 30 min after foot reflexology was done in the intervention group. While in the control group, office BPs were measured at baseline and after resting in a quiet room for 15 and 30 min. A validated, FDA-approved automatic BP device (DINAMAP Pro 300, GE healthcare) with the appropriate cuff size for individual arm circumference was used for measurement. Two BP measurements were taken at 2-min intervals, and the average BP were recorded for analyses.
Change of blood pressure level | Change from Baseline Systolic Blood Pressure at 30 minutes
  The office blood pressures (BP) were measured by a nurse at baseline and at 15 and 30 min after foot reflexology was done in the intervention group. While in the control group, office BPs were measured at baseline and after resting in a quiet room for 15 and 30 min. A validated, FDA-approved automatic BP device (DINAMAP Pro 300, GE healthcare) with the appropriate cuff size for individual arm circumference was used for measurement. Two BP measurements were taken at 2-min intervals, and the average BP were recorded for analyses.
Change of pulse rate | Change from baseline pulse rate at 15 minutes
  The office pulse rate (PR) was measured by a nurse at baseline and at 15 and 30 min after foot reflexology was done in the intervention group. While in the control group, office PR was measured at baseline and after resting in a quiet room for 15 and 30 min.
Change of pulse rate | Change from baseline pulse rate at 30 minutes
  The office pulse rate (PR) was measured by a nurse at baseline and at 15 and 30 min after foot reflexology was done in the intervention group. While in the control group, office PR was measured at baseline and after resting in a quiet room for 15 and 30 min.

SECONDARY OUTCOMES:
Difference in degree of reduction of blood pressure between groups | Difference in degree of reduction of blood pressure from baseline after 30 min
  Compare the degree of reduction of blood pressure between intervention and control group
Difference in degree of reduction of pulse rate between groups | Difference in degree of reduction of pulse rate from baseline after 30 min
  Compare the degree of reduction of pulse rate between intervention and control group

IPD SHARING:
Plan to Share IPD: Yes
Personal contact for IPD
Supporting Information: Study Protocol, SAP
Time Frame: Until 31st December 2020